CLINICAL TRIAL: NCT01587638
Title: Use of Beta-blockers and Risk of New Onset Diabetes
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111198
Record Dates: First submitted 2011-04-14; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension
Keywords: new-onset diabetes; carvedilol; claims analysis; beta-blocker; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Carvedilol; Atenolol; Metoprolol

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hypertensive users of Beta blocker: Patients aged ≥18 years and at least 1 diagnosis of hypertension (ICD-9-CM: 401.xx-405.xx) during this time frame in a US Managed care population
  Interventions: Drug: carvedilol; Drug: cardio selective betablocker

INTERVENTIONS:
Drug: carvedilol — carvedilol immediate-release (IR) and carvedilol controlled-release (CR)
  Other Names: carvedilol immediate-release (IR) and carvedilol controlled-release
Drug: cardio selective betablocker — atenolol, metoprolol succinate, and metoprolol tartrate
  Other Names: atenolol; metoprolol succinate; and metoprolol tartrate

SUMMARY:
This study used an observational, retrospective cohort design to compare the presence and timing of new-onset diabetes (NOD) between hypertensive patients initiating therapy with carvedilol immediate-release (IR) and carvedilol controlled-release (CR) vs the following cardioselective beta blockers (BBs): atenolol, metoprolol succinate, and metoprolol tartrate (referred to hereafter as 'other BB').

The aim of the study was to investigate the likelihood of developing NOD among hypertensive patients initiating carvedilol therapy vs other BB therapy in a real world setting derived from data contained in a large United States (US) managed care database.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a plan captured in the IMS LifeLink Health Plan Claims Database between July 1, 2000 and December 31, 2007
* aged ≥18 years
* at least one pharmacy claim for a beta-blocker of interest (carvedilol immediate-release [IR]/controlled-release [CR], atenolol, metoprolol succinate, or metoprolol tartrate)
* Index date was the first chronologically occurring prescription for any beta-blocker during the enrollment period
* Continuously eligible to receive healthcare services 6 months prior to and 3 months after the index date
* at least 1 diagnosis of hypertension (International Classification of Disease, 9th Revision, Clinical Modification (ICD-9-CM): 401.xx-405.xx) during this time frame.

Exclusion Criteria:

* Diagnosis of diabetes mellitus (ICD-9-CM: 250.xx) and/or a prescription for antidiabetic therapy in the 6 months prior to and/or 3 months after the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective database study identified patients aged ≥18 years with at least one pharmacy claim for a beta-blocker of interest (carvedilol immediate-release [IR]/controlled-release [CR], atenolol, metoprolol succinate, or metoprolol tartrate) identified in the IMS LifeLink Health Plan Claims Database. Index date was the first chronologically occurring prescription for any beta-blocker during the enrollment period (July 1, 2000-December 31, 2007). Patients were identified if they were continuously eligible to receive healthcare services 6 months prior to and 3 months after the index date and at least 1 diagnosis of hypertension (ICD-9-CM: 401.xx-405.xx) during this time frame.
Sampling Method: Non-Probability Sample
Enrollment: 12336 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Rate of New Onset Diabetes (NOD) | From index event (BB prescription) to NOD outcome event (DM diagnosis or antidiabetic Rx) during the effective dates of the database (up to 7 years)
  Rate of NOD per 100 person years. NOD was defined as at least two medical claims with a Diabetes Mellitus diagnosis (ICD-9-CM: 250.xx) or a prescription fill of an antidiabetic medication

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Result] Fonseca V, Sharma PP, Shah M, Deedwania P. Risk of new-onset diabetes mellitus associated with beta-blocker treatment for hypertension. Curr Med Res Opin. 2011 Apr;27(4):799-807. doi: 10.1185/03007995.2011.555477. Epub 2011 Feb 10. PMID 21306286